CLINICAL TRIAL: NCT00660764
Title: Assessment of the Efficacy of Rosuvastatin in Patient Groups With a Dissimilar Risk Profile in an Observational Study (HEROS)
Acronym: HEROS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk - Medical Science Director, AstraZeneca
Other Study IDs: 25V07
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease; Peripheral Vascular Disease; Cerebrovascular Accident; Diabetes
Keywords: cholesterol; coronary heart disease; rosuvastatin; LDL-C goal; hypercholesterolemia; secondary prevention; primary prevention; CVA
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease; Peripheral Vascular Diseases; Stroke; Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients eligible for the study were patients who had not been treated with cholesterol lowering drugs at least in the past three months, with an LDL-C ≥ 3.2 mmol/l. Patients were aged ≥ 18 years and ≤ 70 years (men) and ≤ 75 years (women), according to the advise of the CBO, and could be included in one of the following risk groups: secondary prevention, DM or primary prevention. The general practice investigator made the decision to start treatment with rosuvastatin irrespective of study participation. Patient approved to place anonymous results at the disposal of AstraZeneca
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Oral
  Other Names: Crestor

SUMMARY:
In an observational multi-centre study (HEROS), the effects of starting treatment with rosuvastatin were assessed, on low-density lipoprotein cholesterol (LDL-C) goal achievement, in patients with a dissimilar high-risk profile who had not been treated with cholesterol lowering drugs at least in the past three months. Also set-up costs of rosuvastatin treatment and proportional changes in LDL-C and high-density lipoprotein cholesterol (HDL-C) were studied.

ELIGIBILITY:
Inclusion Criteria:

* patients who had not been treated with cholesterol lowering drugs at least in the past three months, with an LDL-C 3.2 mmol/l.
* According to the advise of the CBO, and could be included in one of the following risk groups: secondary prevention, DM or primary prevention.
* The general practice investigator made the decision to start treatment with rosuvastatin irrespective of study participation.
* Patient approved to place anonymous results at the disposal of AstraZeneca

Exclusion Criteria:

* Patients with symptoms of myalgia, myopathy or liver function insufficiency (including raised serum transaminases) which bear a causal relation to the treatment with statins, patients with familiar dyslipidemia and/or patients with contra-indications for treatment with rosuvastatin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of practices of General Practioners
Sampling Method: Non-Probability Sample
Dates: Start 2003-05; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Effects of starting treatment with rosuvastatin were assessed, on low-density lipoprotein cholesterol (LDL-C) goal achievement, in patients with a dissimilar high-risk profile who hadn't been treated with cholesterol lowering drugs in the past 3 months. | 2 year

SECONDARY OUTCOMES:
Also set-up costs of rosuvastatin treatment and proportional changes in LDL-C and high-density lipoprotein cholesterol (HDL-C) were studied.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid van Geel, Study Chair — CV; Ingeborg Vosjan, Study Chair — CV